CLINICAL TRIAL: NCT02588469
Title: Effects of Exercise and Venous Compression on Upper Airway Resistance in Obese Teenagers With Obstructive Sleep Apnea Syndrome
Brief Title: Exercise and Venous Compression on Upper Airway Resistance in Obese Teenagers With OSA
Acronym: OBESOMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P/2015/250
Record Dates: First submitted 2015-07-22; First posted 2015-10-27 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pediatric Obesity; Sleep Apnea, Obstructive
Keywords: pediatric obesity; obstructive sleep apnea; physical exercise; compression socks; rostral fluid shift
MeSH Terms: conditions — Pediatric Obesity; Sleep Apnea, Obstructive; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional group (Experimental): Physical activity program coupled with compression socks wearing during 3 months.
  Interventions: Other: Interventional group
- control group (Active Comparator): Physical activity program without compression socks during 3 months.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Interventional group — Venous compression leads to beneficial fluid regulation in OSA participants and appears as an efficient tool in OSA management.
  To the investigators knowledge no study assess the impact of the cumulative effect of physical and venous compression program on upper airway resistances in obese teenager with OSA.
  Arms: Interventional group
Other: Control group — Standard obesity care with physical activity program
  Arms: control group

SUMMARY:
The purpose of this study is to assess the effects of physical exercise, associated or not with venous compression of the leg, on obstructive sleep apnea (OSA) severity and upper airway resistance in obese teenagers. Half of the participants will undergo physical exercise and compression socks program, and the other half of subjects will undergo physical exercise program without compression socks.

DETAILED DESCRIPTION:
Obesity is an important factor of OSA development in children and teenagers, and physical activity is a relevant alternative to promote OSA decrease with ou without weight loss.

Physical activity, beyond the improvement of body composition and exercise cardiorespiratory capacity, restricts fluid retaining in the lower limb of the leg by the activation of musculovenous pump. Fluid retaining is involved in OSA severity because of nocturnal fluid shift from legs to rostral zone which promotes pharyngeal oedema development and upper airway collapsibility.

It has been previously shown that venous compression leads to beneficial fluid regulation in OSA subjects and appears as an efficient tool in OSA management.

To the investigators knowledge no study assess the impact of the cumulative effect of physical and venous compression program on upper airway resistances in obese teenager with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescents (BMI > 97th percentile),
* patients aged from 12 to 17 years old, (born between 07/01/2003 and 09/01/1197),
* enrolled in a pediatric obesity center with diet and physical activity programs and psychological management,
* without observed tonsils hypertrophy (Mallampati and Friedman scores),
* without contraindication for bioimpedance analysis, acoustic method and stain gauge plethysmography,
* with physical activity certificate issued by a cardiologist
* covered by the national insurance scheme of his/her legal representative,
* having signed, as well as his(her) legal representative, the informed consent of participation.

Exclusion Criteria:

* Non obese adolescents (BMI < 97th percentile)
* patients aged under 12 or over 17 years old,
* not enrolled in a pediatric obesity center with diet and physical activity programs and psychological management,
* with observed tonsils hypertrophy (Mallampati and Friedman scores),
* with contraindication for bioimpedance analysis, acoustic method and stain gauge plethysmography,
* without physical activity certificate issued by a cardiologist
* uncovered by the national insurance scheme of his/her legal representative,
* not having signed, as well as his(her) legal representative, the informed consent of participation.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Obstructive sleep apnea severity at 3 months. | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Obstructive Sleep Apnea change will be assessed with polysomnography system at baseline and after three months

SECONDARY OUTCOMES:
Upper airway resistances | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  upper airway resistance will be assessed by acoustic method
Fluid shift | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  fluid shift will be assessed by bioimpedance analysis
Calf and neck circumferences | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Calf and neck circumferences will be assessed with nonelastic tape
Calf and neck circumferences | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Calf and neck circumferences will be assessed by plethysmography
Anthropometric parameters | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  weight, height, waist and hip circumferences (body weight scale, standing stadiometer and non-elastic tape)
Body composition | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  fat mass, fat free mass ( by bioimpedance analysis)
Pulmonary function during exercise | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Incremental maximal exercise in cycling ergometer with respiratory gas assessment (metamax)
Metabolic responses | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Glucose, LDL-Cholesterol, HDL-Cholesterol, Total Cholesterol, Triglycerides (ELISA and RIA technics)
Hormonal responses | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  Insulin, leptin, adiponectin, catecholamines (ELISA and RIA technics)
Inflammatory responses | This study includes 2 assessments : baseline (T0) and 3 months (T3)
  C-reactive protein (ELISA and RIA technics)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de soins de suite et de réadaptation La Beline, Salins-les-Bains, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roche J, Corgosinho FC, Damaso AR, Isacco L, Miguet M, Fillon A, Guyon A, Moreira GA, Pradella-Hallinan M, Tufik S, Tulio de Mello M, Gillet V, Pereira B, Duclos M, Boirie Y, Masurier J, Franco P, Thivel D, Mougin F. Sleep-disordered breathing in adolescents with obesity: When does it start to affect cardiometabolic health? Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):683-693. doi: 10.1016/j.numecd.2019.12.003. Epub 2019 Dec 16. PMID 32008915
- [Derived] Roche J, Gillet V, Perret F, Mougin F. Obstructive Sleep Apnea and Sleep Architecture in Adolescents With Severe Obesity: Effects of a 9-Month Lifestyle Modification Program Based on Regular Exercise and a Balanced Diet. J Clin Sleep Med. 2018 Jun 15;14(6):967-976. doi: 10.5664/jcsm.7162. PMID 29852904